CLINICAL TRIAL: NCT05901636
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human Phase 1/2a Study to Evaluate Safety, Reactogenicity and Immunogenicity of a Universal Influenza (Uniflu) Vaccine With INFLUENZA G1 mHA in Healthy Adults
Brief Title: A Clinical Study to Evaluate an Experimental Universal Influenza Vaccine, INFLUENZA G1 mHA, in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CR108777; VAC21148FLZ1001 (Other: Janssen Vaccines & Prevention B.V.); 2019-004635-23 (EudraCT Number)
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Influenza Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- INFLUENZA G1 mHA Dose Level 1 (Experimental): Participants will receive single intramuscular (IM) injection of INFLUENZA G1 mHA Dose level 1 on Days 1 and 57 in Cohort 1.
  Interventions: Biological: INFLUENZA G1 mHA
- INFLUENZA G1 mHA Dose Level 1 along with Al(OH)3 (Experimental): Participants will receive single IM injection of INFLUENZA G1 mHA Dose level 1 with Aluminum Hydroxide (Al[OH])3 adjuvant on Days 1 and 57 in Cohort 1.
  Interventions: Biological: INFLUENZA G1 mHA; Biological: Al(OH)3
- Placebo (Placebo Comparator): Participants will receive IM injection of placebo on Days 1 and 57 in Cohorts 1 and 2.
  Interventions: Biological: Placebo
- INFLUENZA G1 mHA Dose Level 2 (Experimental): Participants will receive single IM injection of INFLUENZA G1 mHA Dose level 2 on Days 1 and 57 in Cohort 2.
  Interventions: Biological: INFLUENZA G1 mHA
- INFLUENZA G1 mHA Dose Level 2 along with Al(OH)3 (Experimental): Participants will receive single IM injection of INFLUENZA G1 mHA Dose level 2 with Al(OH)3 adjuvant on Days 1 and 57 in Cohort 2.
  Interventions: Biological: INFLUENZA G1 mHA; Biological: Al(OH)3
- INFLUENZA G1 mHA Dose Level 2 + Placebo (Experimental): Participants will receive single IM injection of INFLUENZA G1 mHA Dose level 2 on Day 1 and placebo on Day 57 in Cohort 2.
  Interventions: Biological: INFLUENZA G1 mHA
- INFLUENZA G1 mHA Dose Level 2 along with Al(OH)3 + Placebo (Experimental): Participants will receive single IM injection of INFLUENZA G1 mHA Dose level 2 with Al(OH)3 adjuvant on Day 1 and placebo on Day 57 in Cohort 2.
  Interventions: Biological: INFLUENZA G1 mHA; Biological: Al(OH)3

INTERVENTIONS:
Biological: INFLUENZA G1 mHA — INFLUENZA G1 mHA will be administered intramuscularly.
  Arms: INFLUENZA G1 mHA Dose Level 1; INFLUENZA G1 mHA Dose Level 1 along with Al(OH)3; INFLUENZA G1 mHA Dose Level 2; INFLUENZA G1 mHA Dose Level 2 + Placebo; INFLUENZA G1 mHA Dose Level 2 along with Al(OH)3; INFLUENZA G1 mHA Dose Level 2 along with Al(OH)3 + Placebo
Biological: Placebo — Placebo will be administered intramuscularly.
  Arms: Placebo
Biological: Al(OH)3 — Al(OH)3 will be administered intramuscularly.
  Arms: INFLUENZA G1 mHA Dose Level 1 along with Al(OH)3; INFLUENZA G1 mHA Dose Level 2 along with Al(OH)3; INFLUENZA G1 mHA Dose Level 2 along with Al(OH)3 + Placebo

SUMMARY:
The primary purpose of this study is to evaluate safety/ reactogenicity of INFLUENZA G1 mini-hemagglutinin stem-derived protein vaccine antigen (mHA), with or without Al(OH)3 adjuvant, in healthy adults greater than or equal to (>=) 18 to less than or equal to (<=) 45 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy as confirmed by medical history, physical examination, vital signs, and clinical laboratory tests performed at screening
* Contraceptive (birth control) use by female participants should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies. Before randomization, participants who were born female must be either: a) not of childbearing potential; b) of childbearing potential and practicing a highly effective method of contraception and agreeing to remain on such a method of contraception from signing the informed consent until 3 months after the last dose of study vaccine. Use of hormonal contraception should start at least 28 days before the first administration of study vaccine. Highly effective methods for this study include: hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion/ligation procedures, vasectomized partner (the vasectomized partner should be the sole partner for that participant), and sexual abstinence
* All female participants of childbearing potential must: a) have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening; b) have a negative urine beta-hCG pregnancy test immediately prior to each study vaccine administration
* Must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the laboratory screening tests are outside the laboratory normal reference ranges and additionally within the limits of toxicity Grade 2 according to the US FDA toxicity scale the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant and appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Contraindication to IM injections and blood draws, example, bleeding disorders
* Clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius (100.4 degree Fahrenheit) within 24 hours prior to the planned first dose of study vaccine; randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor
* History of severe allergic reaction (for example, anaphylaxis) or other serious adverse reactions to vaccines or vaccine excipients (specifically the excipients of the study vaccine[s])
* Abnormal function of the immune system resulting from: a) clinical conditions (example, autoimmune disease or immunodeficiency) or their treatments expected to have an impact on the immune response elicited by the study vaccine; b) chronic or recurrent use of systemic corticosteroids within 2 months before administration of study vaccine and during the study; c) administration of antineoplastic and immunomodulating agents or radiotherapy expected to have an impact on the immune response elicited by the study vaccine within 6 months before administration of study vaccine and during the study
* History of acute polyneuropathy (example, Guillain-Barré syndrome) or chronic idiopathic demyelinating polyneuropathy
* Received treatment with immunoglobulins (including monoclonal antibodies) expected to impact the vaccine-induced immune response in the 2 months or blood products in the 3 months before the planned administration of the first dose of study vaccine or has any plans to receive such treatment during the study.
* Received an investigational drug or used an invasive investigational medical device within 30 days or received an investigational vaccine within 6 months before the planned administration of the first dose of study vaccine, or received an investigational biological product within 3 months or 5 half-lives, whichever is longer, before the planned study intervention, or is currently enrolled or plans to participate in another investigational study or observational clinical study during the course of this study
* Pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of study vaccine. Oocyte donation is prohibited while enrolled in this study
* Received or plans to receive: licensed live attenuated vaccines - within 28 days before or after planned administration of the first or subsequent study vaccination[s]; other licensed (not live) vaccines (not including seasonal influenza vaccines) - within 14 days before or after planned administration of the first or subsequent study vaccination[s]; seasonal influenza vaccines - within 4 months before planned administration of the first study vaccination until the end of the study (that is, any individual who requires a seasonal influenza vaccination for occupational or other reasons will be excluded)
* Has received a pandemic influenza vaccine (other than Hemagglutinin Type 1 and Neuraminidase Type 1 [H1N1]) in a previous pandemic influenza vaccine study at any time prior to randomization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (4):
- United States (4):
  - Floridian Clinical Research LLC, Miami Lakes, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Clinical Trials Managements, LLC, Metairie, Louisiana
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of 2 Cohorts: Cohort 1 (Group 1 to 3) and Cohort 2 (Group 4 to 8). Participants were enrolled in a staggered approach with safety evaluations (Day 8) in place before extending enrollment in each cohort and progressing from one cohort to the next. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Groups:
- Group 1: Influenza A G1 mHA 45 mcg (Two Doses): Participants received a single dose of 45 micrograms (mcg) Influenza A Group 1 (G1) hemagglutinin stem-derived protein antigen (mHA) vaccine as intramuscular (IM) injection on Day 1 and Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses): Participants received a single dose of 45 mcg Influenza A G1 mHA with Aluminum Hydroxide (Al[OH]3) vaccine as IM injection on Day 1 and Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Group 4: Influenza A G1 mHA 135 mcg (Two Doses): Participants received a single dose of 135 mcg Influenza A G1 mHA vaccine as IM injection on Day 1 and Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses): Participants received a single dose of 135 mcg Influenza A G1 mHA with Al(OH)3 vaccine as IM injection on Day 1 and Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose): Participants received a single dose of 135 mcg Influenza A G1 mHA vaccine as IM injection on Day 1 and a single dose of placebo matching to Influenza A G1 mHA vaccine on Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose): Participants received a single dose of 135 mcg Influenza A G1 mHA with Al(OH)3 vaccine as IM injection on Day 1 and a single dose of placebo matching to Influenza A G1 mHA vaccine on Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Group 3 and Group 8: Placebo (Two Doses): Participants received a single dose of placebo matching to Influenza A G1 mHA vaccine as IM injection on Day 1 and Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
Period: Overall Study
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Started | 25 | 25 | 25 | 25 | 25 | 25 | 20
Number of Participants Who Received Vaccination 1 | 25 | 25 | 25 | 25 | 25 | 25 | 20
Number of Participants Who Received Vaccination 2 | 24 | 23 | 23 | 25 | 23 | 24 | 20
Number of Participants Who Received 2 Doses of Placebo in Group 3 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Number of Participants Who Received 2 Doses of Placebo in Group 8 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Completed | 24 | 23 | 22 | 22 | 23 | 21 | 17
Not Completed | 1 | 2 | 3 | 3 | 2 | 4 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 1 | 3 | 1
Not completed — Non- Compliance With Study Schedule | 0 | 0 | 2 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Influenza A G1 mHA 45 mcg (Two Doses): Participants received a single dose of 45 mcg Influenza A G1 mHA vaccine as IM injection on Day 1 and Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses): Participants received a single dose of 45 mcg Influenza A G1 mHA with Al(OH)3 vaccine as IM injection on Day 1 and Day 57. Participants were followed up for safety for a minimum period of 28 days after each vaccination (up to Day 29 and Day 85 respectively) and for long term safety until 1 year after the first vaccination (Day 365).
- Total: Total of all reporting groups
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses) | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20 | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.6 (7.77) | 31.2 (8.31) | 34.3 (7.13) | 35.1 (7.22) | 32.0 (7.06) | 32.5 (7.96) | 31.6 (7.69) | 32.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15 | 18 | 13 | 16 | 12 | 89
  Male | 17 | 18 | 10 | 7 | 12 | 9 | 8 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 12 | 11 | 12 | 7 | 9 | 68
  Not Hispanic or Latino | 19 | 14 | 13 | 14 | 13 | 18 | 11 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 9 | 6 | 5 | 5 | 5 | 5 | 3 | 38
  White | 15 | 18 | 19 | 20 | 20 | 20 | 17 | 129
  More than one race | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 25 | 25 | 25 | 25 | 20 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) Within 7 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited local AEs were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site) AEs for which participants were specifically questioned and which were noted by participants in a diary for 7 days post vaccination (day of vaccination and the subsequent 7 days). Solicited local AEs included injection site pain/tenderness, erythema, and swelling at the vaccination site.
Time Frame: Within 7 Days after vaccination 1 on Day 1 (from Day 1 up to Day 8)
Population: Full analysis set (FAS) included all participants with at least 1 vaccination documented. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 5 | 12 | 3 | 13 | 6 | 14 | 1

2. Primary Outcome: Number of Participants With Solicited Local AEs Within 7 Days After Vaccination 2
Description: as for outcome 1
Time Frame: Within 7 Days after vaccination 2 on Day 57 (from Day 57 up to Day 64)
Population: FAS included all participants with at least 1 vaccination documented. Here 'N' (overall number of participants analyzed) refers to the number of participants who received vaccination 2. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 5 | 9 | 5 | 8 | 2 | 5 | 2

3. Primary Outcome: Number of Participants With Worst Grade (at Least Grade 3) Solicited Local AEs Within 7 Days After Vaccination 1
Description: AE: any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. AE does not necessarily have a causal relationship with intervention. Solicited local AEs used to assess reactogenicity of vaccine. Pre-defined local AEs (pain/tenderness, erythema and swelling at injection site) were noted by participants in a diary for 7 days post vaccination (day of vaccination and subsequent 7 days). Severity was assessed using food and drug administration (FDA) toxicity grading scale- Pain: Grade (G) 1 (mild; does not interfere with activity); G2 (moderate; requires modification in activity/use of medications); G3 (severe; inability to do usual activities/use of narcotic pain reliever); G4 (life threatening; hospitalization), Erythema and swelling: G 1 (mild; 25 -50 millimeter [mm]); G2 (moderate; 51 -100 mm); G3 (severe; greater than [>] 100 mm); G4 (life threatening; hospitalization/necrosis or exfoliative dermatitis).
Time Frame: Within 7 Days after vaccination 1 on Day 1 (from Day 1 up to Day 8)
Population: FAS included all participants with at least 1 vaccination documented. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Worst Grade (at Least Grade 3) Solicited Local AEs Within 7 Days After Vaccination 2
Description: AE: any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. AE does not necessarily have a causal relationship with intervention. Solicited local AEs used to assess reactogenicity of vaccine. Pre-defined local AEs (pain/tenderness, erythema and swelling at injection site) were noted by participants in a diary for 7 days post vaccination (day of vaccination and subsequent 7 days). Severity was assessed using FDA toxicity grading scale- Pain: Grade 1 (mild; does not interfere with activity); Grade 2 (moderate; requires modification in activity/use of medications); Grade 3 (severe; inability to do usual activities/use of narcotic pain reliever); Grade 4 (life threatening; hospitalization), Erythema and swelling: Grade 1 (mild; 25 -50 mm); Grade 2 (moderate; 51 -100 mm); Grade 3 (severe; >100 mm); Grade 4 (life threatening; hospitalization/necrosis or exfoliative dermatitis).
Time Frame: Within 7 Days after vaccination 2 on Day 57 (from Day 57 up to Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Duration of Solicited Local AEs That Occurred Within 7 Days After Vaccination 1
Description: Duration of solicited AEs was defined as number of days from the start of the event until resolution of the event. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited local AEs were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site) AEs for which participants were specifically questioned and which were noted by participants in a diary for 7 days post vaccination (day of vaccination and the subsequent 7 days). Solicited local AEs included injection site pain/tenderness, erythema, and swelling at the vaccination site.
Time Frame: From Day 1 up to Day 365
Population: FAS included all participants with at least 1 vaccination documented. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for specified rows. n=0 indicated that no participant experienced the specified AE in respective arm. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Measure: Median (Full Range); unit: Days
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 5 | 12 | 3 | 13 | 6 | 14 | 1
Days
  Vaccination site erythema: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 2 | 0
  Vaccination site erythema | 1.0 [1 to 1] | 1.0 [1 to 1] | 1.0 [1 to 1] |  |  | 1.0 [1 to 1] |
  Vaccination site swelling: number analyzed (Participants) | 1 | 2 | 1 | 0 | 0 | 0 | 0
  Vaccination site swelling | 1.0 [1 to 1] | 1.0 [1 to 1] | 5.0 [5 to 5] |  |  |  |
  Vaccination site pain: number analyzed (Participants) | 5 | 12 | 2 | 13 | 6 | 14 | 1
  Vaccination site pain | 1.0 [1 to 2] | 2.5 [1 to 7] | 4.0 [3 to 5] | 2.0 [1 to 4] | 1.0 [1 to 1] | 2.0 [1 to 7] | 3.0 [3 to 3]

6. Primary Outcome: Duration of Solicited Local AEs That Occurred Within 7 Days After Vaccination 2
Description: as for outcome 5
Time Frame: From Day 57 up to Day 365
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 5 | 9 | 5 | 8 | 2 | 5 | 2
Days
  Vaccination site erythema: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Vaccination site erythema |  |  |  |  |  |  | 1.0 [1 to 1]
  Vaccination site swelling: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Vaccination site swelling |  |  |  |  |  |  | 1.0 [1 to 1]
  Vaccination site pain | 1.0 [1 to 2] | 2.0 [1 to 6] | 2.0 [1 to 4] | 1.5 [1 to 3] | 1.0 [1 to 1] | 1.0 [1 to 2] | 1.0 [1 to 1]

7. Primary Outcome: Number of Participants With Solicited Systemic AEs Within 7 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited systemic AEs were used to assess the reactogenicity of the study vaccine. Systemic events (fatigue, headache, nausea, myalgia, and fever) for which participants were specifically questioned, and which were noted by participants in a diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Within 7 Days after vaccination 1 on Day 1 (from Day 1 up to Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 7 | 12 | 6 | 9 | 7 | 12 | 4

8. Primary Outcome: Number of Participants With Solicited Systemic AE Within 7 Days After Vaccination 2
Description: as for outcome 7
Time Frame: Within 7 Days after vaccination 2 on Day 57 (from Day 57 up to Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 4 | 8 | 7 | 9 | 6 | 8 | 4

9. Primary Outcome: Number of Participants With Worst Grade (at Least Grade 3) Solicited Systemic AEs Within 7 Days After Vaccination 1
Description: AE was any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. AE does not necessarily have causal relationship with intervention. Solicited systemic AEs used to assess reactogenicity of vaccine. Systemic events (fatigue, headache, nausea, myalgia, fever) for which participants were specifically questioned and were noted by participants in a diary for 7 days post vaccination (day of vaccination and subsequent 7 days). Severity assessed by FDA toxicity grading scale- Fever: Grade (G) 1 (mild; 38.0-38.4 degrees Celsius [C]), G2 (moderate; 38.5-38.9 degrees C), G3 (severe; 39.0-40.0 degrees C), G4 (>40.0 degrees C); fatigue, headache, nausea and myalgia: G1 (mild; does not interfere with activity), G2 (moderate; requires modification in activity/use of medications), G3 (severe; inability to do usual activities/use of medications); G4 (life threatening; hospitalization).
Time Frame: Within 7 Days after vaccination 1 on Day 1 (from Day 1 up to Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Worst Grade (at Least Grade 3) Solicited Systemic AE Within 7 Days After Vaccination 2
Description: as for outcome 9
Time Frame: Within 7 Days after vaccination 2 on Day 57 (from Day 57 up to Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 0 | 0 | 0 | 1 | 1 | 0 | 0

11. Primary Outcome: Duration of Solicited Systemic AEs That Occurred Within 7 Days After Vaccination 1
Description: Duration of solicited AEs was defined as number of days from the start of the event until resolution of the event. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited systemic AEs were used to assess the reactogenicity of the study vaccine. Systemic events (fatigue, headache, nausea, myalgia, and fever) for which participants were specifically questioned, and which were noted by participants in a diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: From Day 1 up to Day 365
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 7 | 12 | 6 | 9 | 7 | 12 | 4
Days
  Fatigue: number analyzed (Participants) | 6 | 7 | 6 | 5 | 6 | 8 | 3
  Fatigue | 2.0 [1 to 7] | 3.0 [1 to 6] | 1.5 [1 to 3] | 1 [1 to 1] | 1.5 [1 to 5] | 4.5 [1 to 8] | 1.0 [1 to 7]
  Headache: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 8 | 0
  Headache | 3.0 [2 to 4] | 4.0 [1 to 6] | 1.5 [1 to 2] | 1.0 [1 to 1] | 5.5 [4 to 7] | 4.5 [1 to 6] |
  Nausea: number analyzed (Participants) | 2 | 2 | 2 | 0 | 4 | 3 | 0
  Nausea | 1.0 [1 to 1] | 1.0 [1 to 1] | 1.0 [1 to 1] |  | 1.0 [1 to 1] | 5.0 [2 to 7] |
  Myalgia: number analyzed (Participants) | 4 | 8 | 3 | 4 | 2 | 8 | 1
  Myalgia | 1.0 [1 to 2] | 3.0 [1 to 6] | 1.0 [1 to 5] | 1.0 [1 to 2] | 3.5 [1 to 6] | 1.0 [1 to 5] | 1.0 [1 to 1]
  Pyrexia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Duration of Solicited Systemic AEs That Occurred Within 7 Days After Vaccination 2
Description: as for outcome 11
Time Frame: From Day 57 up to Day 365
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 4 | 8 | 7 | 9 | 6 | 8 | 4
Days
  Fatigue: number analyzed (Participants) | 3 | 4 | 5 | 6 | 5 | 7 | 3
  Fatigue | 6.0 [2 to 15] | 6.0 [4 to 8] | 1.0 [1 to 5] | 1.0 [1 to 9] | 1.0 [1 to 4] | 4.0 [1 to 7] | 1.0 [1 to 2]
  Headache: number analyzed (Participants) | 2 | 4 | 4 | 3 | 2 | 7 | 1
  Headache | 9.0 [1 to 17] | 5.0 [1 to 8] | 3.0 [2 to 6] | 3.0 [2 to 7] | 2.0 [2 to 2] | 4.0 [1 to 7] | 2.0 [2 to 2]
  Nausea: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 2 | 2
  Nausea | 1.0 [1 to 1] |  |  | 1.0 [1 to 1] |  | 3.5 [1 to 6] | 1.5 [1 to 2]
  Myalgia: number analyzed (Participants) | 2 | 6 | 3 | 2 | 0 | 5 | 0
  Myalgia | 1.5 [1 to 2] | 2.5 [1 to 5] | 2.0 [1 to 3] | 2.0 [1 to 3] |  | 1.0 [1 to 6] |
  Pyrexia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Pyrexia |  |  |  |  |  |  | 8.0 [8 to 8]

13. Primary Outcome: Number of Participants With Solicited Systemic AEs Related to Study Vaccine Within 7 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited systemic AEs were used to assess the reactogenicity of the study vaccine. Systemic events (fatigue, headache, nausea, myalgia, and fever) for which participants were specifically questioned, and which were noted by participants in a diary for 7 days post vaccination (day of vaccination and the subsequent 7 days). Number of participants with solicited systemic AEs related to study vaccine were reported.
Time Frame: Within 7 Days after vaccination 1 on Day 1 (from Day 1 up to Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 7 | 12 | 6 | 9 | 7 | 12 | 4

14. Primary Outcome: Number of Participants With Solicited Systemic AEs Related to Study Vaccine Within 7 Days After Vaccination 2
Description: as for outcome 13
Time Frame: Within 7 Days after vaccination 2 on Day 57 (from Day 57 up to Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 4 | 8 | 7 | 9 | 6 | 8 | 3

15. Primary Outcome: Number of Participants With Unsolicited AEs Within 28 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have causal relationship with intervention. An unsolicited AE was defined as all AEs for which the participants were not specifically questioned in the participant's reactogenicity diary.
Time Frame: Within 28 Days after vaccination 1 on Day 1 (from Day 1 up to Day 29)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 1 | 1 | 0 | 1 | 0 | 1 | 1

16. Primary Outcome: Number of Participants With Unsolicited AEs Within 28 Days After Vaccination 2
Description: as for outcome 15
Time Frame: Within 28 Days after vaccination 2 on Day 57 (from Day 57 up to Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 1 | 1 | 2 | 3 | 2 | 2 | 1

17. Primary Outcome: Number of Participants With Worst Grade (At Least Grade 3) Unsolicited AEs Within 28 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have causal relationship with intervention. An unsolicited AE was defined as all AEs for which the participants were not specifically questioned in the participant's reactogenicity diary. The severity of AEs was assessed by FDA toxicity grading scale: Grade 1 (mild; symptoms causing no or minimal interference with usual social and functional activities); Grade 2 (moderate; symptoms causing greater than minimal interference with usual social and functional activities; Grade 3 (severe; symptoms causing inability to perform usual social and functional activities and requires medical intervention); Grade 4 (life threatening; hospitalization).
Time Frame: Within 28 Days after vaccination 1 on Day 1 (from Day 1 up to Day 29)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Worst Grade (At Least Grade 3) Unsolicited AEs Within 28 Days After Vaccination 2
Description: as for outcome 17
Time Frame: Within 28 Days after vaccination 2 on Day 57 (from Day 57 up to Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 0 | 0 | 0 | 1 | 1 | 0 | 0

19. Primary Outcome: Duration of Unsolicited AEs That Occurred Within 28 Days After Vaccination 1
Description: Duration of unsolicited AEs was defined as number of days from the start of the event until resolution of the event. An AE was any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have causal relationship with intervention. An unsolicited AE was defined as all AEs for which the participants were not specifically questioned in the participant's reactogenicity diary. Unsolicited AEs that occurred within 28 days after vaccination 1 are reported below.
Time Frame: From Day 1 up to Day 365
Population: FAS: all participants with at least 1 vaccination documented. N=number of participants evaluable for this outcome measure; n (number analyzed)=number of participants evaluable for specified rows. N=0 indicated that data was not collected and analyzed as no participant experienced any AE in specified arm. n=0 indicated that no participant experienced the specified AE in respective arm. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Measure: Median (Full Range); unit: Days
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 1
Days
  Anaemia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Anaemia |  |  |  |  |  |  | 57.0 [57 to 57]
  Dermatitis contact: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Dermatitis contact |  |  |  |  |  | 11.0 [11 to 11] |
  Diarrhoea: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Diarrhoea |  | 1.0 [1 to 1] |  |  |  |  |
  Nasopharyngitis: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Nasopharyngitis | 11.0 [11 to 11] |  |  |  |  |  |
  Ventricular extrasystoles: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ventricular extrasystoles |  |  |  | 1.0 [1 to 1] |  |  |

20. Primary Outcome: Duration of Unsolicited AEs That Occurred Within 28 Days After Vaccination 2
Description: Duration of unsolicited AEs was defined as number of days from the start of the event until resolution of the event. An AE was any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have causal relationship with intervention. An unsolicited AE was defined as all AEs for which the participants were not specifically questioned in the participant's reactogenicity diary. Unsolicited AEs that occurred within 28 days after vaccination 2 are reported below.
Time Frame: From Day 57 up to Day 365
Population: FAS included all participants with at least 1 vaccination documented. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for specified rows. n=0 indicates that no participant experienced the specified AE in respective arm. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Measure: Median (Full Range); unit: Days
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 2 | 2 | 1
Days
  Anaemia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Anaemia |  |  |  |  | 34.0 [34 to 34] |  |
  Arthralgia: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Arthralgia |  | 3.0 [3 to 3] |  |  |  |  |
  Blood pressure increased: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood pressure increased |  |  |  | 20.0 [20 to 20] |  |  |
  Gastroenteritis: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Gastroenteritis |  |  |  | 7.0 [7 to 7] |  |  |
  Hypertension: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypertension |  |  |  | 252.0 [252 to 252] |  |  |
  Influenza like illness: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 1 | 0
  Influenza like illness |  |  | 6.0 [6 to 6] | 7.0 [7 to 7] | 4.0 [4 to 4] | 7.0 [7 to 7] |
  Leukopenia: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Leukopenia |  |  | 52.0 [52 to 52] |  |  |  |
  Nephrolithiasis: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Nephrolithiasis | 14.0 [14 to 14] |  |  |  |  |  |
  Otitis media acute: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Otitis media acute |  |  |  | 7.0 [7 to 7] |  |  |
  Pulmonary embolism: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Pulmonary embolism |  |  |  |  |  |  | 92.0 [92 to 92]
  Rhinorrhoea: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Rhinorrhoea |  |  |  | 2.0 [2 to 2] |  |  |
  Sinusitis: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Sinusitis |  |  |  |  |  | 8.0 [8 to 8] |
  Transient ischaemic attack: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Transient ischaemic attack |  |  |  | 3.0 [3 to 3] |  |  |

21. Primary Outcome: Number of Participants With Unsolicited AEs Related to Study Vaccine Within 28 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have causal relationship with intervention. An unsolicited AE was defined as all AEs for which the participants were not specifically questioned in the participant's reactogenicity diary. Number of participants with any unsolicited AEs related to study vaccine were reported.
Time Frame: Within 28 Days after vaccination 1 on Day 1 (from Day 1 up to Day 29)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Number of Participants With Unsolicited AEs Related to Study Vaccine Within 28 Days After Vaccination 2
Description: as for outcome 21
Time Frame: Within 28 Days after vaccination 2 on Day 57 (from Day 57 up to Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 23 | 23 | 25 | 23 | 24 | 20
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and SAEs Related to Study Vaccine
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Serious AE was the AE resulting in any of following outcomes/deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants with SAEs and SAEs related to study vaccine were reported.
Time Frame: From first vaccination (Day 1) up to Day 365
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25 | 20
Participants
  SAE | 0 | 0 | 0 | 2 | 0 | 0 | 0
  SAE related to study vaccine | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Geometric Mean Concentration of Antibodies Binding to Hemagglutinin (HA) Stem or Full-length HA Protein as Measured by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: Geometric mean concentration of antibodies binding to HA stem or full-length HA protein as measured by ELISA (H5-ELISA and mHA ELISA) was reported. HA stem derived protein vaccine antigen (mHA) derived from H1N1 A/California/07/2009 virus strain. Per-protocol Immunogenicity population was denoted as PPI. As planned, combined data was collected and analyzed for participants who received Placebo in Groups 3 and 8.
Time Frame: Days 29 and 85
Population: PPI included all randomized and vaccinated participants for whom immunogenicity data were available excluding samples taken on or after the date when a participant experiences a major protocol deviation expected to impact the immunogenicity outcomes. 'n' (number analyzed)=number of participants evaluable for specified rows. n=0 indicates that no participant was available for the analysis in the respective arm for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Unit per milliliter (EU)/mL
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
Number analyzed (Participants) | 24 | 25 | 25 | 25 | 25 | 25 | 20
ELISA Unit per milliliter (EU)/mL
  H5 A/Vietnam/1203/2004 ELISA: Day 29: number analyzed (Participants) | 23 | 25 | 22 | 24 | 24 | 24 | 20
  H5 A/Vietnam/1203/2004 ELISA: Day 29 | 2919 [1563 to 5450] | 2990 [1970 to 4538] | 3240 [1750 to 5998] | 4468 [2659 to 7507] | 3998 [2262 to 7068] | 5468 [3429 to 8717] | 329 [197 to 549]
  H5 A/Vietnam/1203/2004 ELISA: Day 85: number analyzed (Participants) | 22 | 23 | 21 | 22 | 20 | 24 | 20
  H5 A/Vietnam/1203/2004 ELISA: Day 85 | 3015 [1738 to 5233] | 2892 [1879 to 4450] | 3413 [1984 to 5870] | 4276 [2755 to 6638] | 3044 [1774 to 5224] | 3087 [1955 to 4874] | 363 [228 to 578]
  H1 mHA A/California/07/2009 ELISA: Day 29: number analyzed (Participants) | 23 | 25 | 22 | 24 | 24 | 24 | 20
  H1 mHA A/California/07/2009 ELISA: Day 29 | 27285 [16056 to 46368] | 28343 [20284 to 39604] | 31894 [17465 to 58242] | 43631 [28230 to 67437] | 44575 [28632 to 69397] | 57306 [41346 to 79426] | 3337 [2109 to 5280]
  H1 mHA A/California/07/2009 ELISA: Day 85: number analyzed (Participants) | 22 | 23 | 21 | 22 | 20 | 24 | 20
  H1 mHA A/California/07/2009 ELISA: Day 85 | 28875 [18668 to 44665] | 29496 [21477 to 40509] | 36459 [23450 to 56686] | 45667 [33342 to 62547] | 31845 [20601 to 49224] | 32809 [24239 to 44409] | 3383 [2136 to 5358]

ADVERSE EVENTS:
Time Frame: All cause mortality: From baseline (pre-vaccination Day 1) up to Day 365; SAE: From the day of vaccination 1 (Day 1) up to Day 365; Other AEs: Solicited AEs: within 7 days after vaccination 1 on Day 1 (up to Day 8), within 7 days after vaccination 2 on Day 57 (up to Day 64); Unsolicited AEs: within 28 days after vaccination 1 on Day 1 (up to Day 29 ), within 28 days after vaccination 2 on Day 57 (up to Day 85)
Description: All Cause Mortality: All randomized participants. SAE and Other AEs: FAS included all participants with at least 1 vaccination documented.
Arm/Group | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) | Group 3 and Group 8: Placebo (Two Doses)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25 | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 2/25 | 0/25 | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 9/25 | 16/25 | 8/25 | 18/25 | 9/25 | 16/25 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) (N=25) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) (N=25) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) (N=25) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) (N=25) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) (N=25) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) (N=25) | Group 3 and Group 8: Placebo (Two Doses) (N=20)
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Influenza A G1 mHA 45 mcg (Two Doses) (N=25) | Group 2: Influenza A G1 mHA 45 mcg With Al(OH)3 (Two Doses) (N=25) | Group 4: Influenza A G1 mHA 135 mcg (Two Doses) (N=25) | Group 5: Influenza A G1 mHA 135 mcg With Al(OH)3 (Two Doses) (N=25) | Group 6: Influenza A G1 mHA 135 mcg (First Dose) + Placebo (Second Dose) (N=25) | Group 7: Influenza A G1 mHA 135 mcg With Al(OH)3 (First Dose) + Placebo (Second Dose) (N=25) | Group 3 and Group 8: Placebo (Two Doses) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Solicited) (Gastrointestinal disorders) | 3 | 2 | 2 | 1 | 4 | 3 | 2
Fatigue (Solicited) (General disorders) | 8 | 8 | 7 | 10 | 7 | 8 | 5
Pyrexia (Solicited) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination Site Erythema (Solicited) (General disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 1
Vaccination Site Pain (Solicited) (General disorders) | 7 | 13 | 5 | 14 | 7 | 15 | 3
Vaccination Site Swelling (Solicited) (General disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 5 | 10 | 4 | 5 | 2 | 10 | 1
Headache (Solicited) (Nervous system disorders) | 3 | 7 | 5 | 6 | 3 | 9 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT05901636/Prot_001.pdf
  • Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT05901636/SAP_002.pdf